CLINICAL TRIAL: NCT06078228
Title: Assessment of Ultrasonographic Carotid Artery Corrected Flow Time and Internal Jugular Vein Collapsibility Index in Prediction of Hypotension During Induction of General Anesthesia
Brief Title: Prediction of Hypotension During Induction of General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD205/2023
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Propofol - Fentanyl- Atracurium — investigate the reliability of preanesthetic ultrasound measurements of the carotid artery FTc and the internal jugular vein collapsibility index in predicting hypotension during the induction of general anesthesia.
  Other Names: Atropine

SUMMARY:
Post induction hypotension is closely related to postoperative complications. Patients are at high risk of hypotension due to preexisting hypovolemia and the vasodilatory effects of induction agents. Ultrasonographic measurement of the Carotid artery corrected flow time and internal jugular vein collapsibility index may predict post induction hypotension.

DETAILED DESCRIPTION:
* Type of Study: Observational Prospective Cohort Design.
* Study Setting and ethical consideration: The approval of the Scientific Research Ethics Committee of the Faculty of Medicine, Ain Shams University will be obtained before starting work on the study. This study will be conducted in operating theatres of Ain Shams University Hospitals. Informed written consents to participate will be obtained from the patients.
* Study Period: One year (October 2023-October 2024)
* Study Population: Adult patient undergoing elective surgeries.

ELIGIBILITY:
Inclusion Criteria:

* 1- Patients of American Society of Anesthesiologists (ASA) physical status I to II of both genders.

  2- Aged 18-65 years. 3- Elective surgeries under general anesthesia. 4- BMI less than 40.

Exclusion Criteria:

* Patients with

  1. Renal diseases.
  2. Hepatic diseases.
  3. ASA scores of 3-4.
  4. The presence of a left ventricular ejection fraction less than 50%.
  5. Age under 18 years old.
  6. Patient refusal.
  7. Coronary heart disease.
  8. Cardiac disease including cardiomyopathy and mild to severe valve disease.
  9. Pulmonary hypertension.
  10. Peripheral arterial disease.
  11. Preoperative cervical vascular ultrasound abnormalities including plaque, stenosis and anatomical variation.
  12. Any previous neck surgery or trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patient undergoing elective surgeries.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-08-17 (Estimated); Study Completion 2024-08-17 (Estimated)

PRIMARY OUTCOMES:
the predictive value of the carotid Ftc for prediction of hypotension. | one year
  to investigate the reliability of preanesthetic ultrasound measurements of the carotid artery FTc and the internal jugular vein collapsibility index in predicting hypotension during the induction of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marina George, MD candidate, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT06078228/Prot_000.pdf
  • Informed Consent Form (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT06078228/ICF_001.pdf